CLINICAL TRIAL: NCT00932087
Title: Characterization of Low Density Lipoprotein and Mechanism of the Pro Aggregant Effect Through Oxidant Stress and Lipid Exchange
Acronym: ECLIPSE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Philippe MOULIN, MD PhD, Hospices Civils de Lyon
Other Study IDs: 2008.516
Record Dates: First submitted 2009-06-22; First posted 2009-07-02 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes; Metabolic Syndrome
Keywords: Platelet function; diabetes; metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- type 2 diabetics with metabolic syndrome
  Interventions: Procedure: Blood sample
- metabolic syndrome without diabetes
  Interventions: Procedure: Blood sample
- type 1 diabetes
  Interventions: Procedure: Blood sample
- control
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample for lipidomic study

SUMMARY:
Case control design: lipidomic study in 12 type 2 diabetics with metabolic syndrome, 12 metabolic syndrome without diabetes, 12 subjects with type 1 diabetes and 12 controls

ELIGIBILITY:
Inclusion Criteria:

* statin and fibrate Wash out for one week
* HbA1c>7% and <12% (Arms 1 and 3)
* HbA1c<6% (Arms 2 and 4)
* Metabolic sd according NCEP III (3 out 4 criteria) (Arms 1 and 2)

Exclusion Criteria:

* secondary CV prevention

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group 1: type 2 diabetics with metabolic syndrome group 2: metabolic syndrome without diabetes group 3: subjects with type 1 diabetes group 4: controls
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Level of plasma isoprostane and lipoperoxides | at baseline

SECONDARY OUTCOMES:
TXA2 and PF4 levels after platelet activation of control platelet exposed to LDL | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOULIN, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Fédération d'Endocrinologie-Diabétologie-Maladies métaboliques-Nutrition - Hôpital Cardiovasculaire et Pneumologique, Lyon, France

REFERENCES:
- [Derived] Colas R, Sassolas A, Guichardant M, Cugnet-Anceau C, Moret M, Moulin P, Lagarde M, Calzada C. LDL from obese patients with the metabolic syndrome show increased lipid peroxidation and activate platelets. Diabetologia. 2011 Nov;54(11):2931-40. doi: 10.1007/s00125-011-2272-8. Epub 2011 Aug 17. PMID 21847583